CLINICAL TRIAL: NCT05291442
Title: Improving Resilience and Quality of Life of Stroke Patients: A Mixed Method Study
Brief Title: Improving Resilience and Quality of Life of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CS1-21079
Record Dates: First submitted 2022-03-18; First posted 2022-03-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stroke Patient; Caregiver
Keywords: Resilience; Family system nursing; Self-efficacy; Quality of life; Complexity science; Transition theory; Caregiver; Stroke.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: To integrate Family System Care and Theme Care Action Module to improve resilience, family function, self-efficacy, and quality of life for stroke patients and their caregivers.
  First, understand the care needs of patients and caregivers, and apply The Specific Thematic Nursing Care Action Modules (STNC-AM) platform for education and training.
  The Specific Thematic Nursing Care Action Modules (STNC-AM) platform that we present here is an educational program that integrates education and coaching. STNC-AM has six key aspects: stroke prevention, management of emotions, management of fatigue, physical activity, caregiver training, and integrative resources. Each scope contains detailed care guidance.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group received no intervention, except for the regular care followed by the nurses in general in the rehabilitation ward.
- Intervention group (Experimental): To integrate Family System Care and Theme Care Action Module to improve resilience, family function, self-efficacy, and quality of life for stroke patients and their caregivers.
  First, understand the care needs of patients and caregivers, and apply The Specific Thematic Nursing Care Action Modules (STNC-AM) platform for education and training.
  The Specific Thematic Nursing Care Action Modules (STNC-AM) platform that we present here is an educational program that integrates education and coaching. STNC-AM has six key aspects: stroke prevention, management of emotions, management of fatigue, physical activity, caregiver training, and integrative resources. Each scope contains detailed care guidance.
  Interventions: Other: To integrate Family System Care and Theme Care Action Module

INTERVENTIONS:
Other: To integrate Family System Care and Theme Care Action Module — First, understand the care needs of patients and caregivers, and apply The Specific Thematic Nursing Care Action Modules (STNC-AM) platform for education and training.
  The Specific Thematic Nursing Care Action Modules (STNC-AM) platform that we present here is an educational program that integrates education and coaching. STNC-AM has six key aspects: stroke prevention, management of emotions, management of fatigue, physical activity, caregiver training, and integrative resources. Each scope contains detailed care guidance.
  Arms: Intervention group

SUMMARY:
This study aims to (1) test the effect of Family System Care and Theme Care Action Module on resilience, family function, self-efficacy, and quality of life for stroke patients and their families and caregivers; and (2) interview stroke survivors (experimental group) using a semi-structured questionnaire to achieve a mix of qualitative and quantitative methodologies.

DETAILED DESCRIPTION:
A randomized control-group pretest-posttest design was adopted. We also used a semi-structured questionnaire to qualitatively interview stroke survivors. The National Institute of Health Stroke Scale (NIHSS), Chronic Disease Self-Efficacy scales, Resilience Scale, McMaster Family Assessment Device, and Quality of Life Scale were used to test the intervention effects. Further, complex scientific concepts will be used to analyze the transition experience of stroke survivors.

Expected outcomes: The Family System Care and Theme Care Action Module can improve family function, resilience, self-efficacy, and quality of life for stroke patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

stroke patient:

* Those who can use language expression, over 20 years old.
* Within 1-6 months of new onset; (c) Patients willing to participate. Family caregivers
* family members or relatives and friends over 20 years of age who provide the care recipients' personal needs, financial, psychological, emotional care, etc.

Exclusion Criteria:

* Aphasia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
resilience_change is being assessed | 3rd day after admission (T1). 2-3 weeks after admission (Time 2). 2-3 days before discharge (Time 3).
  Investigators use the Resilience Scale to evaluate the resilience for stroke patients. Total scores ranged from 25 to 175, with higher scores as indicating greater resilience.
family function_change is being assessed | 3rd day after admission (T1). 2-3 weeks after admission (Time 2). 2-3 days before discharge (Time 3).
  Investigators use the McMaster family assessment device to evaluate the family function for stroke patients and their caregiver. Total scores ranged from 12 to 48, with higher scores as indicating greater family function.
self-efficacy_change is being assessed | 3rd day after admission (T1). 2-3 weeks after admission (Time 2). 2-3 days before discharge (Time 3).
  Investigators use the Chronic Disease Self-efficacy Scale to evaluate the self-efficacy for stroke patients. Total scores ranged from 6 to 60, with higher scores as indicating greater self-efficacy.
quality of life_change is being assessed | 3rd day after admission (T1). 2-3 weeks after admission (Time 2). 2-3 days before discharge (Time 3).
  Investigators use the SF-12 Health Survey Version 2(SF-12v2) to evaluate the quality of life for stroke patients and their caregiver. Total scores ranged from 0 to 100, with higher scores as indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Chu Pai, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan